CLINICAL TRIAL: NCT00907582
Title: Autologous Hematopoietic Cell Transplantation for Acute Promyelocytic Leukemia After Relapse With Idarubicin and Busulfan Conditioning
Brief Title: ASCT for Relapsed APL After Molecular Remission
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow recruitment
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Jiong HU, Head, Blood and Marrow Transplantation Center, Rui Jin Hospital, Shanghai Jiao Tong University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MHOPES-APL09
Record Dates: First submitted 2009-05-21; First posted 2009-05-22 (Estimated); Last update posted 2014-12-02 (Estimated); Status verified 2014-11

CONDITIONS: Acute Promyelocytic Leukemia; Relapse
Keywords: PCR negative
MeSH Terms: conditions — Leukemia, Promyelocytic, Acute; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- ASCT in relapsed APL (Experimental): autologous hematopoietic cell transplantation for patients with relapsed APL after achieving molecular remission
  Interventions: Procedure: autologous hematopoietic cell transplantation

INTERVENTIONS:
Procedure: autologous hematopoietic cell transplantation — Autologous hematopoietic cell transplantation and condition with the following:
  idarubicin 15mg/m2•d day -11 and -10; busulfan 0.8mg/kg•q6h day -6 to -3.

SUMMARY:
For relapsed acute promyelocytic leukemia after all-trans retinoic acid (ATRA) and arsenic treatment, remission can be achieved by chemotherapy with ATRA and/or arsenic and addition of mylotarg. Autologous hematopoietic cell transplantation using a polymerase chain reaction (PCR) negative graft is important treatment option to obtain sustainable remission. This study is to test the efficacy and the safety of conditioning regimen with idarubicin and busulfan for relapsed Acute Promyelocytic Leukemia (APL).

DETAILED DESCRIPTION:
Once relapsed acute promyelocytic leukemia achieved molecular remission after all-trans retinoic acid (ATRA) and arsenic treatment, PBSC was mobilized and collected with further confirmation of molecular remission via RT-PCR.

Patients received autologous hematopoietic cell transplantation.

ELIGIBILITY:
Inclusion Criteria:

* Men or women between age 18-60 years old
* Acute promyelocytic leukemia after relapse with confirmed cytogenetics t(15;17) and molecular analysis (PML-RARalpha)
* Mobilized peripheral CD34+ over 2x106/kg with negative PML-RAR alpha confirmed by PCR
* European Cooperative Oncology Group performance status 0-3
* Serum bilirubin < 1.5x the upper limit of normal (ULN)
* Serum alanine transaminase (ALT)/aspartate transaminase values < 2.5 x ULN
* Subjects (or their legally acceptable representatives) must signed an informed consent document indicating that they understanding the purpose of and procedures required for the study and are willing to participate in the study

Exclusion Criteria:

* Woman of child bearing potential
* Serum creatinine > 400 Micromol/l after initial resuscitation patients with previous Grade 2-4 peripheral neuropathy
* Uncontrolled diabetes (if receiving antidiabetic agents, subjects must be on a stable dose for at least 3 months before first dose of study drug)
* Uncontrolled or severe cardiovascular disease including myocardial infarction within 6 months of enrollment, uncontrolled angina, clinically significant pericardial disease, or III-IV heart failure
* Known allergy to idarubicin

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 5 (Actual)
Dates: Start 2009-06; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
disease free survival | 3 years

SECONDARY OUTCOMES:
overall survival | 3 years
transplantation related mortality | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: JIong HU, M.D., Principal Investigator — Shanghai Rui Jin Hospital
Locations (1):
- Rui Jin Hospital, Shanghai JiaoTong University School of Medicine, Shanghai, China